CLINICAL TRIAL: NCT02505412
Title: Prevalence of Subtle Myocardial Deformation Abnormalities in Asymptomatic Nf-1 Patients: is Cardiac Screening Needed?
Brief Title: Subtle Myocardial Deformation Abnormalities in Asymptomatic Nf-1 Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, michal roll (telavivsmo), Tel-Aviv Sourasky Medical Center
Other Study IDs: TLV-0212-15
Record Dates: First submitted 2015-07-16; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Subtle myocardial deformation abnormalities in asymptomatic nf-1 patients: is cardiac screening needed?

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic NF1 patients
* aged 0-17y and 11 months

Exclusion Criteria:

* clinical heart failure,
* history of cardiovascular disease
* chronic renal insufficiency

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Consecutive asymptomatic NF1 patients, aged 0-17y and 11 month, who will visit the investigators' Neurofibromatosis tertiary outpatients clinics
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
myocardial deformation indices as measured in percentage (change of original length) | up to 2 years